CLINICAL TRIAL: NCT02395653
Title: An Open Label Evaluation of the Safety and Clinical Utility of the Active, Separated System With Enhanced Controller (SSEC) Fentanyl 40 mcg for the Management of Acute Postoperative Pain in Pediatric Patients 12 to Less Than 18 Years of Age
Brief Title: Safety and Clinical Utility Study of SSEC Fentanyl 40 mcg for Acute Post-op Pain Management in Pediatric Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Collaborators: Incline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PD2013-002; 2014-002405-37 (EudraCT Number)
Record Dates: First submitted 2015-03-10; First posted 2015-03-23 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-09

CONDITIONS: Pain, Postoperative
Keywords: Pediatric; Postoperative; Pain Management
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SSEC Fentanyl (Experimental): SSEC fentanyl iontophoretic transdermal system, 40 mcg fentanyl per activation.
  Interventions: Drug: fentanyl

INTERVENTIONS:
Drug: fentanyl — An opioid that has been administered parenterally as an anesthetic and analgesic for more than 20 years.
  Other Names: IONSYS

SUMMARY:
The objective of this study is to evaluate the safety and clinical utility of the active, SSEC fentanyl 40 micrograms (mcg) for the management of acute, postoperative pain in pediatric participants.

DETAILED DESCRIPTION:
An open label evaluation of the safety and clinical utility of the active, SSEC fentanyl 40 mcg for the management of acute postoperative pain in pediatric participants 12 to less than 18 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Participants whose parent(s) or guardian(s) have/has signed and dated an informed consent form for the participant to participate in the study, or participants who have provided written assent to participate in the study
* Male or female inpatients, age 12 to <18 years of age inclusive on the day of surgery
* Participants capable of understanding and cooperating with the requirements of the study, including being able to report their pain intensity using the 11-point Numeric Rating Scale and operate the SSEC
* American Society of Anesthesiologists physical status I, II or III
* Body weight of at least 40.0 kilogram (kg)
* Postoperative participants who have undergone general or regional anesthesia for abdominal, pelvic/genitourinary, orthopedic, or thoracic surgery
* Postoperative participants who have been observed during recovery and are expected to remain hospitalized and have pain requiring parenteral opioids (that is, intravenous [IV] patient-controlled anesthesia) for the next 24 hours or longer
* Participants who are awake and breathing spontaneously with a respiratory rate of 14 to 18 breaths per minute, peripheral capillary oxygen saturation ≥93% (with or without supplemental oxygen), and able to answer questions and follow commands
* Participants who have been observed during recovery, who are awake, able to answer questions and follow commands, and who have been comfortable for at least 30 minutes, with a pain intensity score ≤4 (numeric rating scale 0-10), with or without titration to comfort with IV opioids

Exclusion Criteria:

* Participants who have undergone any surgery on the airway, head, or neck
* Participants who received an extended-release opioid within 48 hours prior to Hour 0 or who are expected to have postoperative analgesia supplied by a continuous regional technique or participant-controlled epidural analgesia
* Participants with a history of allergy or hypersensitivity to fentanyl, skin adhesives, and/or cetylpyridinium chloride
* Participants who are expected to require intensive care or will likely require additional surgical procedures within 36 hours
* Participants who received intra-operative and/or postoperative administration of opioids other than morphine, hydromorphone, fentanyl, sufentanil, or alfentanil. Exception: If there are no medical contraindications, meperidine (pethidine) up to 0.5 milligram/kg IV is permitted during recovery for shivering
* Participants who require airway support (nasal or oropharyngeal airway intubation, or laryngeal mask airway at the time of final baseline assessments (that is, at the time of IONSYS application [Hour 0])
* Participants who are known or suspected to be opioid tolerant, have a history of opioid dependence within 3 months before the start of the study, or who are known to have used illicit drugs or alcohol within 14 days of the start of the study
* Participants with active generalized skin disorders or active local skin disease that precludes SSEC application to the chest or upper arm
* Participants with any coexisting major medical conditions that are likely to interfere with study procedures including, but not limited to, psychiatric conditions, chronic depression, suicidal ideation, autism
* Positive pregnancy test for any female

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2016-09-12 (Actual); Study Completion 2016-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot J Krane, MD, Principal Investigator — Stanford Children's Health
Locations (10):
- United States (10):
  - Packard Children's Hospital at Stanford, Palo Alto, California
  - University of Miami/Jackson Memorial Hospital, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Johns Hopkins Hospital, Charlotte R. Bloomberg Children's Center, Baltimore, Maryland
  - St. Louis Children's Hospital, St Louis, Missouri
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Children's Medical Center of Dallas, Dallas, Texas
  - Harborview Medical Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Chelly JE, Grass J, Houseman TW, Minkowitz H, Pue A. The safety and efficacy of a fentanyl patient-controlled transdermal system for acute postoperative analgesia: a multicenter, placebo-controlled trial. Anesth Analg. 2004 Feb;98(2):427-433. doi: 10.1213/01.ANE.0000093314.13848.7E. PMID 14742382
- [Background] Grond S, Hall J, Spacek A, Hoppenbrouwers M, Richarz U, Bonnet F. Iontophoretic transdermal system using fentanyl compared with patient-controlled intravenous analgesia using morphine for postoperative pain management. Br J Anaesth. 2007 Jun;98(6):806-15. doi: 10.1093/bja/aem102. PMID 17519263
- [Background] Hartrick CT, Bourne MH, Gargiulo K, Damaraju CV, Vallow S, Hewitt DJ. Fentanyl iontophoretic transdermal system for acute-pain management after orthopedic surgery: a comparative study with morphine intravenous patient-controlled analgesia. Reg Anesth Pain Med. 2006 Nov-Dec;31(6):546-54. doi: 10.1016/j.rapm.2006.08.011. PMID 17138198
- [Background] Minkowitz HS, Rathmell JP, Vallow S, Gargiulo K, Damaraju CV, Hewitt DJ. Efficacy and safety of the fentanyl iontophoretic transdermal system (ITS) and intravenous patient-controlled analgesia (IV PCA) with morphine for pain management following abdominal or pelvic surgery. Pain Med. 2007 Nov-Dec;8(8):657-68. doi: 10.1111/j.1526-4637.2006.00257.x. PMID 18028044
- [Background] Minkowitz HS, Yarmush J, Donnell MT, Tonner PH, Damaraju CV, Skowronski RJ. Safety and tolerability of fentanyl iontophoretic transdermal system: findings from a pooled data analysis of four clinical trials. J Opioid Manag. 2010 May-Jun;6(3):203-10. doi: 10.5055/jom.2010.0018. PMID 20642249
- [Background] Viscusi ER, Reynolds L, Chung F, Atkinson LE, Khanna S. Patient-controlled transdermal fentanyl hydrochloride vs intravenous morphine pump for postoperative pain: a randomized controlled trial. JAMA. 2004 Mar 17;291(11):1333-41. doi: 10.1001/jama.291.11.1333. PMID 15026400
- [Background] Viscusi ER, Reynolds L, Tait S, Melson T, Atkinson LE. An iontophoretic fentanyl patient-activated analgesic delivery system for postoperative pain: a double-blind, placebo-controlled trial. Anesth Analg. 2006 Jan;102(1):188-94. doi: 10.1213/01.ane.0000183649.58483.77. PMID 16368828
- [Background] Viscusi ER, Siccardi M, Damaraju CV, Hewitt DJ, Kershaw P. The safety and efficacy of fentanyl iontophoretic transdermal system compared with morphine intravenous patient-controlled analgesia for postoperative pain management: an analysis of pooled data from three randomized, active-controlled clinical studies. Anesth Analg. 2007 Nov;105(5):1428-36, table of contents. doi: 10.1213/01.ane.0000281913.28623.fd. PMID 17959978

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric participants from 12 to less than 18 years of age who had undergone general or regional anesthesia for elective abdominal, pelvic/genitourinary, orthopedic, or thoracic surgery.
Pre-assignment Details: Screening within 3 weeks of study start included review of inclusion/exclusion criteria, informed consent signature, medical history, height, weight, vital signs, American Society of Anesthesiologists physical status, and a review of the Separated System With Enhanced Controller (SSEC) for delivery of 40 micrograms (mcg) fentanyl/dose.
Groups:
- SSEC Fentanyl: Post-surgery, participants received fentanyl via the active IONSYS® SSEC fentanyl iontophoretic transdermal system that provided on-demand systemic delivery of 40 mcg fentanyl per dose for up to 24 hours, or a maximum of 80 doses, whichever came first, for up to 3 consecutive days (up to 72 hours).
Period: Overall Study
Arm/Group | SSEC Fentanyl
Started | 71
Received at Least 1 Dose of Study Drug (Participants included in the Safety Population.) | 61
Completed | 59
Not Completed | 12
Not completed — Exclusion Criteria Met at Screening | 4
Not completed — Consent Withdrawn at Screening | 1
Not completed — SSEC Application But With 0 Dose | 1
Not completed — Investigator Decision at Screening | 1
Not completed — Inclusion Criteria Not Met at Screening | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population included all participants who received ≥1 dose of fentanyl from the SSEC.
Arm/Group | SSEC Fentanyl
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.7 (1.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Assessment Of Participant's Ability To Use The SSEC
Description: Investigator's assessment of participant's ability to use the SSEC system safely and effectively. The assessment consisted of a 4-level categorical evaluation (poor, fair, good, and excellent). Because of the descriptive nature of this study, no formal statistical hypothesis testing was performed.
Time Frame: Completed at the time of the participant's termination of study treatment (up to 72 hours after study drug administration)
Population: The Evaluable Population consists of all participants who received fentanyl from the SSEC for at least 3 hours.
Measure: Number; unit: participants
Arm/Group | SSEC Fentanyl
Number analyzed (Participants) | 61
participants
  Poor | 1
  Fair | 2
  Good | 10
  Excellent | 48
  Missing | 0

2. Primary Outcome: Assessment Of Adherence Of The SSEC System To Skin
Description: The adhesion of each SSEC was evaluated immediately prior to removal at each 24-hour time point, or at early withdrawal. Adhesion was recorded using the following classification: System adhered to at least 90% of the application area with no edges unattached; System adhered between 75% and 89%; System was <75% adhered and not taped; System was secured with tape. The number of SSEC systems for all time points in each category is presented. Because of the descriptive nature of this study, no formal statistical hypothesis testing was performed.
Time Frame: Immediately prior to removal at each 24-hour time point, or at early withdrawal, for up to 3 consecutive days (up to 72 hours)
Population: The Evaluable Population consists of all participants who received fentanyl from the SSEC for at least 3 hours.
Measure: Number; unit: SSEC systems
Units Other Than Participants: SSEC systems used by 61 participants
Arm/Group | SSEC Fentanyl
Number analyzed (Participants) | 61
Number analyzed (SSEC systems used by 61 participants) | 107
SSEC systems
  ≥90% of area with no edges unattached | 97
  75% to 89% | 6
  <75% adhered and not taped | 3
  System was secured with tape | 1
  Not assessed | 0

3. Secondary Outcome: Change From Baseline To 1 Hour And 24 Hours In Skin Irritation Score After SSEC Removal
Description: Skin irritation at the SSEC application site was to be assessed immediately prior to placement of the study system and at 1 and 24 hours after removal of each study system. The application site was to be scored using the following scale: 0=No evidence of irritation; 1=Minimal erythema, barely perceptible; 2=Definite erythema, readily visible, minimal edema, or minimal papular response; 3=Erythema and papules; 4=Definite edema; 5=Erythema, edema, and papules; 6=Vesicular eruption; 7=Strong reaction spreading beyond the application site.
Time Frame: Baseline, 1 hour and 24 hours after SSEC removal.
Population: The Evaluable Population consists of all participants who received fentanyl from the SSEC for at least 3 hours.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SSEC Fentanyl
Number analyzed (Participants) | 61
units on a scale
  System 1, Hour 1 | 1.1 (0.94)
  System 1, Hour 24: number analyzed (Participants) | 48
  System 1, Hour 24 | 1.8 (1.43)
  System 2, Hour 1: number analyzed (Participants) | 39
  System 2, Hour 1 | 1.0 (0.61)
  System 2, Hour 24: number analyzed (Participants) | 34
  System 2, Hour 24 | 1.6 (1.33)
  System 3, Hour 1: number analyzed (Participants) | 5
  System 3, Hour 1 | 1.0 (1.22)
  System 3, Hour 24: number analyzed (Participants) | 4
  System 3, Hour 24 | 0.8 (1.26)

4. Secondary Outcome: Number Of Participants To Experience Clinically Relevant Respiratory Depression (CRRD)
Description: Respiratory function and occurrence of CRRD was defined as simultaneous occurrence of bradypnoea (respiratory rate <10 breaths per minute for participants 9-15 years of age and sustained for 1 minute, or <8 breaths per minute for participants 16-17 years of age), with excessive sedation (that is, the participant is not easily aroused).
Time Frame: From the time of application of the first system through 7 days following end of study drug administration.
Population: The Evaluable Population consists of all participants who received fentanyl from the SSEC for at least 3 hours.
Measure: Number; unit: participants
Arm/Group | SSEC Fentanyl
Number analyzed (Participants) | 61
participants
  Bradypnoea | 0
  Excessive Sedation | 0
  Simultaneous Bradypnoea and Excessive Sedation | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of application of the first system through 7 days following the end of study drug administration.
Arm/Group | SSEC Fentanyl
All-Cause Mortality (participants affected / at risk) | 0/61
Serious Adverse Events (participants affected / at risk) | 1/61
Other Adverse Events (participants affected / at risk) | 44/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSEC Fentanyl (N=61)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SSEC Fentanyl (N=61)
Dizziness (Nervous system disorders) | 7 (9)
Application site erythema (General disorders) | 10 (10)
Application site papules (General disorders) | 10 (10)
Pyrexia (General disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 19 (23)
Nausea (Gastrointestinal disorders) | 18 (19)
Constipation (Gastrointestinal disorders) | 11 (11)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No